CLINICAL TRIAL: NCT02992730
Title: Predictors of Adjuvant Endocrine Therapy in Women With Breast Cancer
Acronym: WHIP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: Sheppard_WHIP_Study
Record Dates: First submitted 2016-12-05; First posted 2016-12-14 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer Female
Keywords: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva Sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women Diagnosed with Breast Cancer: Observational - Usual Care
  Interventions: Behavioral: No Intervention

INTERVENTIONS:
Behavioral: No Intervention — No Intervention

SUMMARY:
Breast cancer is the leading cancer diagnosed in women and the second cause of cancer death. Of all racial/ethnic groups in the US, Black women have the highest rate of breast cancer deaths. Two-thirds of Black breast cancer patients have estrogen receptor (ER) positive tumors that can be treated with adjuvant hormonal therapy. If taken for the full five years, this therapy has been shown to reduce mortality by 50%. However, ER positive Black women are more likely to die from their breast cancer as ER positive White women. Preliminary data suggest that non-adherence to adjuvant hormonal therapy could explain some of this disparity. To date, no study has systematically examined psychosocial, healthcare, and biological factors that predict adherence to hormonal therapy in Black women with breast cancer. To begin to fill this knowledge gap, Investigators will conduct a prospective cohort study of 422 ER positive Black breast cancer patients recruited from health maintenance organizations (HMOs). Our primary outcome is adherence to therapy at 36 months post initiation. Specific aims are to: 1) Examine psychosocial factors (e.g. health beliefs, socio-cultural values, etc.) that predict adherence to hormonal therapy; 2) Identify clinical (e.g., side effects), and biological (e.g., stage, etc.) factors that predict adherence to hormonal therapy; and 3) Evaluate healthcare variables (e.g., communication, management of side effects, etc.) that predict adherence. Investigators will also explore the role of CYP2D6 genetic variations in adherence to hormonal therapy which is novel and will increase knowledge about this genetic factor in Blacks. The study is focused on the time-period (first 3 years) when women appear to be the most vulnerable to terminating treatment prematurely. A better understanding of predictors of adherence in Black women may help target interventions and ultimately improve potentially avoidable adverse breast cancer outcomes in this underserved group.

DETAILED DESCRIPTION:
Investigators will employ the Adherence Model of Behavior to identify clinical, psychosocial, and healthcare delivery predictors of longitudinal hormonal therapy adherence in women with (hormone receptor) HR positive breast cancer. This study is significant because: (1) most breast cancers in Blacks and Whites are HR positive (~75%)1,27; (2) hormonal therapy is recommend for all women with HR positive cancer since it reduces recurrence and mortality; (3) women who adhere to hormonal therapy have lower mortality than those who do not28; (4) adherence to hormonal therapy is suboptimal, even in HMO settings; (5) current guidelines recommend at least 5 years of hormonal therapy6; (6) along with Whites, investigators will examine adherence behaviors in Blacks, a group reported to have poorer outcomes than Whites, even among HR positive cases of similar stage;) past studies have documented poor adherence but few have systematically examined reasons for non-adherence. Overall, our results will be clinically useful and will inform interventions and pharmacogenetics research. For instance, if investigators find that communication strongly influences adherence, investigators can develop and implement patient self-efficacy or physician reminder-based interventions to enhance communication about adherence between patients and clinicians in HMOs. If investigators find that different factors predict adherence in Blacks versus Whites, investigators can develop tailored interventions. The PI has extensive experience developing tailored interventions to improve communication and uptake of chemotherapy in Blacks and Latinas.The next sections highlight the background that supports the significance of our research.

ELIGIBILITY:
Inclusion Criteria:

* Non-recurrent invasive breast cancer (AJCC Stages I-IV)
* Any race
* English or Spanish speaking and/or reading
* Initiated hormonal therapy within 12 months of definitive diagnosis

Exclusion Criteria:

* HR Negative
* Under the age of 21
* Non-English or Spanish Speaking

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants for this study are ER positive women over the age of 21 diagnosed with breast cancer.
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2011-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to hormonal therapy at 36 months post initiation - Survey | Baseline to end of followup - 3 years.
  Examine psychosocial factors (e.g. health beliefs, socio-cultural values, etc.) that predict adherence to hormonal therapy.
  Evaluate healthcare variables (e.g., communication, management of side effects, etc.) that predict adherence.

SECONDARY OUTCOMES:
Clinical Factors - Medical Record Review | Baseline to the end of follow-up - 3 years.
  Identify clinical (e.g., side effects), and biological (e.g., stage, etc.) factors that predict adherence to hormonal therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edmonds MC, Sutton AL, Cummings Y, Sheppard VB. Opportunities to Improve Women's Health: Engaging Racial/Ethnic Diverse Women to Provide Biospecimens for Research. J Womens Health (Larchmt). 2021 Sep;30(9):1321-1327. doi: 10.1089/jwh.2020.8502. Epub 2021 Jan 11. PMID 33428522